CLINICAL TRIAL: NCT00918554
Title: Corticosteroid Sparing Effect of Methotrexate in Patients With Sarcoid- Associated Uveitis: A Double Blind, Randomized, Placebo Controlled-study -UVEXATE
Brief Title: Efficacy Study of Methotrexate to Treat Sarcoid-associated Uveitis
Acronym: UVEXATE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient number of inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P070140
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2013-06

CONDITIONS: Sarcoid-associated Uveitis; Ocular Sarcoidosis; Macular Edema
Keywords: Sarcoid-associated uveitis; Macular oedema; Methotrexate; Conventional corticosteroids sparing agent.
MeSH Terms: conditions — Macular Edema | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methotrexate (Experimental)
  Interventions: Drug: Methotrexate
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — All patients will receive three pulses of methylprednisolone (5 mg/kg) followed by four weeks of prednisone (1 mg/kg daily). After randomization, patients will receive either prednisone (1 mg/kg daily) plus methotrexate (0.3 mg/kg weekly) or prednisone (1 mg/kg daily) plus placebo. Therapies will be administered orally. Corticosteroids will be progressively tapered when macular oedema completely resolve. Unilateral macular oedema relapses will be treated with a single local injection triamcinolone acetonide. Increasing dose of prednisone will be administered in case of bilateral macular oedema relapses.
  Arms: Methotrexate
Drug: Placebo — All patients will receive three pulses of methylprednisolone (5 mg/kg) followed by four weeks of prednisone (1 mg/kg daily). After randomization, patients will receive either prednisone (1 mg/kg daily) plus methotrexate (0.3 mg/kg weekly) or prednisone (1 mg/kg daily) plus placebo. Therapies will be administered orally. Corticosteroids will be progressively tapered when macular oedema completely resolve. Unilateral macular oedema relapses will be treated with a single local injection of triamcinolone acetonide. Increasing dose of prednisone will be administered in case of bilateral macular oedema relapses.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether methotrexate is a effective corticosteroid sparing agent in the treatment of sarcoid-associated uveitis.

DETAILED DESCRIPTION:
Macular oedema remains a significant cause of blindness. Corticosteroids are effective in the treatment of sarcoid-associated macular oedema but more than 50% of relapses occur when corticosteroids are tapered. Methotrexate (MTX) at low dose has been shown to be an effective and safe steroid-sparing agent for lung sarcoidosis and compilation of reported small series of patients with sarcoid-associated uveitis suggest that only 25% of relapses could be achieved with low dose MTX. We decide therefore to test the clinical efficacy of MTX in sarcoid-associated uveitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Provided written consent for participation in the trial prior to any study-specific procedures or requirements
* Posterior uveitis or panuveitis associated with macular oedema defined as increased macular thickness (more than 250 mm assessed by Stratus TD-OCT or 300 mm with Cirrus SD-OCT ) and/or the presence of cystoid spaces in the macula, and the absence of epiretinal membranes.
* Patient with oral contraception
* Posterior uveitis or panuveitis associated with macular oedema
* Patients with histologically proven sarcoidosis or a presumed sarcoidosis. In case of a non caseating granuloma in biopsy tissues, the patients with presumed sarcoidosis meet at least 2 of the 4 following criteria: typical changes on chest radiography and computed tomography; predominantly CD4 lymphocytosis in bronchoalveolar lavage (BAL) fluid; elevated serum ACE levels; elevated gallium or 5 fluorodeoxyglucose uptake

Exclusion Criteria:

* Patients who do not fulfill the inclusion criteria
* Other causes of uveitis
* Extra ophthalmologic manifestations of sarcoidosis justifying corticosteroids
* Patients previously treated with immunosuppressive agents or corticosteroids of more than 10 mg daily over 15 days.
* Patients with life-threatening conditions
* Chronic hepatopathy or renal failure
* Uncontrolled diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Percentage of macular oedema relapses. Every two weeks for five months, the amount of macular oedema will be assessed by Optical Coherence Tomography. | at 26 weeks

SECONDARY OUTCOMES:
Cumulated dose of prednisone | at 26 weeks
Number of triamcinolone injections | at 26 weeks
Adverse effects | at 26 weeks
Percentage of patients with best corrected visual acuity under 0.1, 0.2 and 0. | at 26 weeks
Percentage of patients with active anterior and /or posterior uveitis | at 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien ABAD, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital Avicenne - Service de Médecine Interne, Bobigny
  - CHU Michallon de Grenoble, Grenoble